CLINICAL TRIAL: NCT06832436
Title: Assessment of Left And Right Atrial Strain in Septic Shock
Brief Title: Atrial Strain in Septic Shock
Acronym: ALARMS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Henri Mondor University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PI2025_843_0034
Record Dates: First submitted 2025-02-11; First posted 2025-02-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Septic Shock; Left Atrial Strain; Right Atrial Strain; Transthoracic Echocardiography; Speckle Tracking; Echocardiographic Software; Reproducibility; Critical Care
Keywords: transthoracic echocardiography; septic shock; left atrial strain; right atrial strain; speckle tracking; echocardiographic software; AutoStrain; Bland-Altman analysis; reproducibility; critical care
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Septic shock is a critical condition associated with high mortality. Transthoracic echocardiography is widely used to evaluate cardiac function and guide treatment. Left and right atrial strain (LAS and RAS) measured via speckle tracking echocardiography have shown prognostic value in cardiovascular diseases. However, differences exist between echocardiographic software, leading to challenges in result comparability. This study aims to compare LAS and RAS measurements between ECHOPAC and UWS software, evaluate AutoStrain technology, and assess reproducibility across observers. The study is non-interventional and will use retrospective echocardiographic data from patients treated for septic shock. The findings will contribute to improving measurement standardization in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: >18 years
* Adult patients admitted to critical care for septic shock (SEPSIS-3 definition)
* TTE performed as part of medical management
* No objection to data usage

Exclusion Criteria:

* Pregnancy
* Moderate to severe valvular regurgitation/stenosis (>grade 2)
* Ventricular or supraventricular tachyarrhythmia (HR >140 bpm) at the time of TTE
* Poor echogenicity preventing LAS measurement
* Mechanical circulatory support
* Pacemaker dependence
* Patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to critical care for septic shock (SEPSIS-3 definition)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
variation of LASr between ECOPAC and UWS | 1 year
  Agreement of LAS Reservoir Phase (LASr) measurement in manual mode between ECHOPAC and UWS

SECONDARY OUTCOMES:
variation of LAScd between ECHOPAC and UWS | 1 year
  Comparison of LAS Conduit (LAScd) measurements in manual mode between ECHOPAC and UWS
variation of LASct between ECHOPAC and UWS | 1 year
  Comparison of LAS Conduit (LAScd) and Contraction (LASct) measurements in manual mode between ECHOPAC and UWS
Comparison of LASr measurements in apical 2-chamber views | 1 year
  Comparison of LASr measurements in apical 2-chamber views in manual mode between ECHOPAC and UWS
Comparison of LAScd measurements in apical 2-chamber views | 1 year
  Comparison of LAScd measurements in apical 2-chamber views in manual mode between ECHOPAC and UWS
Comparison of LASct measurements in apical 2-chamber views | 1 year
  Comparison of LASct measurements in apical 2-chamber views in manual mode between ECHOPAC and UWS
Comparison of right atrial strain RASr between ECHOPAC and UWS | 1 year
  Comparison of right atrial strain (RASr) in manual mode between ECHOPAC and UWS
Comparison of right atrial strain RAScd between ECHOPAC and UWS | 1 year
  Comparison of right atrial strain RAScd in manual mode between ECHOPAC and UWS
Comparison of right atrial strain RASct between ECHOPAC and UWS | 1 year
  Comparison of right atrial strain RASct in manual mode between ECHOPAC and UWS
Comparison of LAS in AutoStrain versus manual mode | 1 year
  Comparison of LAS measurements in AutoStrain versus manual mode on UWS
Comparison of RAS in AutoStrain versus manual mode | 1 year
  Comparison of RAS measurements in AutoStrain versus manual mode on UWS
Comparison of LAS measurements in AutoStrain (UWS) versus manual mode on ECHOPAC | 1 year
  Comparison of LAS measurements in AutoStrain (UWS) versus manual mode on ECHOPAC
Comparison of RAS measurements in AutoStrain (UWS) versus manual mode on ECHOPAC | 1 year
  Comparison of RAS measurements in AutoStrain (UWS) versus manual mode on ECHOPAC
Assessment of differences in LAS measurements at end-diastole between ECHOPAC and UWS | 1 year
  Assessment of differences in LAS phase measurements between ECHOPAC and UWS
Assessment of differences in LAS measurements at pre-A between ECHOPAC and UWS | 1 year
  Assessment of differences in LAS measurements at pre-A between ECHOPAC and UWS
Assessment of differences in RAS measurements at end-diastole between ECHOPAC and UWS | 1 year
  Assessment of differences in RAS measurements at end-diastole between ECHOPAC and UWS
Assessment of differences in RAS measurements at pre-A between between ECHOPAC and UWS | 1 year
  Assessment of differences in RAS measurements at pre-A between between ECHOPAC and UWS
Inter-observer reproducibility assessment of manual measurements (UWS and GE) in a sample of 10 patients | 1 year
  Inter-observer reproducibility assessment of manual measurements (UWS and GE) in a sample of 10 patients
Intra-observer reproducibility assessment of manual measurements (UWS and GE) in a sample of 10 patients | 1 year
  Intra-observer reproducibility assessment of manual measurements (UWS and GE) in a sample of 10 patients
Inter-observer reproducibility assessment of AutoStrain measurements (UWS and GE) in a sample of 10 patients | 1 year
  Inter-observer reproducibility assessment of AutoStrain measurements (UWS and GE) in a sample of 10 patients
Intra-observer reproducibility assessment of AutoStrain measurements (UWS and GE) in a sample of 10 patients | 1 year
  Intra-observer reproducibility assessment of AutoStrain measurements (UWS and GE) in a sample of 10 patients

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Salouël, France

IPD SHARING:
Plan to Share IPD: No